CLINICAL TRIAL: NCT07320157
Title: "Women's HPV Education and Its Effects on Knowledge Levels, HPV Screening Behaviors, and HPV Vaccination Uptake: An Interventional Education Study"
Brief Title: The Effect of HPV Education Provided to Women on Their Knowledge Levels, HPV Screening, and Vaccination Uptake
Acronym: HPV-Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Gizem Bilmez, Principal Investigator, Ufuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E-81182178-605-56406
Record Dates: First submitted 2025-12-19; First posted 2026-01-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: HPV (Human Papillomavirus)-Associated; HPV Immunization Status
Keywords: HPV; WOMEN; HEALTH; VACCİNE
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Education Intervention Group (Experimental): An online training session will be scheduled for the intervention group. The training will consist of two 40-minute session. After the online training, the training materials will be shared with the group. One week after the training, an informational brochure prepared on the topic will be sent to the intervention group via WhatsApp as a reminder, and any questions they may have will be answered. Two weeks after delivering the brochure, the questionnaire/scale forms will be administered to both groups as the first follow-up. Eight weeks after the first follow-up, the same forms will be administered again as the post-test. The WhatsApp group will remain open and interaction will be allowed throughout the research period.
  Interventions: Behavioral: Online Education Intervention Group; Other: Contral Group

INTERVENTIONS:
Behavioral: Online Education Intervention Group — An online training session will be scheduled for the intervention group. The training will consist of two 40-minute session. After the online training, the training materials will be shared with the group. One week after the training, an informational brochure prepared on the topic will be sent to the intervention group via WhatsApp as a reminder, and any questions they may have will be answered. Two weeks after delivering the brochure, the questionnaire/scale forms will be administered to both groups as the first follow-up. Eight weeks after the first follow-up, the same forms will be administered again as the post-test. The WhatsApp group will remain open and interaction will be allowed throughout the research period.
Other: Contral Group — No intervention will be applied to the control group. Following the completion of the study, the brochure prepared on the topic will be sent to them via WhatsApp.

SUMMARY:
Type of Study: This study was planned to be an observational study.

Purpose of the Study: To evaluate the impact of HPV education given to women on their knowledge levels and HPV screening and vaccination.The main question[s] it aims to answer [is/are]:

H1: There is a difference in the mean Human Papillomavirus (HPV) Knowledge Scale score between the intervention group women who participated in Human Papillomavirus (HPV) education and the control group women.

H2: There is a difference between the intervention group women and the control group women in terms of their participation in HPV screening tests.

H2: There is a difference between the intervention group women and the control group women in terms of their HPV vaccination status.

Participants Participants will be assigned to a control and intervention group. Online training will be provided to the intervention group, and the results of the training will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Being female
* Women aged 18-35 years
* Ability to speak and understand Turkish at a level sufficient to communicate with the researcher
* Having the technical equipment necessary to participate in a video interview
* No diagnosis of HPV positivity
* Not having received the HPV vaccine
* Not having undergone HPV DNA/Pap smear testing in the past 5 years
* No diagnosis of cervical cancer
* Voluntary willingness to participate in the study
* No diagnosis of a psychiatric disorder

Exclusion Criteria:

* Being male
* Having severe physical or cognitive impairments that prevent completing the questionnaire
* Being under 18 years of age or over 35 years of age
* Inability to speak or understand Turkish
* Lack of technical equipment to participate in a video interview
* Having a diagnosis of HPV positivity
* Having received the HPV vaccine
* Having undergone HPV DNA/Pap smear testing in the past 5 years
* Having a diagnosis of cervical cancer
* Having a diagnosed psychiatric disorder

Not agreeing to participate in the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Because the study evaluates an intervention related to cervical health, only female participants will be included.
Enrollment: 64 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Change in HPV Knowledge Score | Baseline (before intervention), 2 weeks after brochure delivery (first follow-up), and 8 weeks after the first follow-up (final follow-up)
  Change in participants' HPV Knowledge Scale scores measured at baseline, first follow-up, and final follow-up. The measure evaluates the effect of the online education and brochure intervention compared to the control group.

SECONDARY OUTCOMES:
Sustained HPV Knowledge Score (Knowledge Retention) | Knowledge retention will be assessed by comparing HPV Knowledge Scale scores between groups at the final follow-up. Higher scores indicate better long-term retention of information provided by the intervention.
  Final follow-up (8 weeks after the first follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- UfUk UNİVERSİTY, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to privacy and confidentiality concerns of the participants, individual participant data will not be shared.